CLINICAL TRIAL: NCT03201081
Title: Impact of a Motivational Resistance-training Program on Adherence and Body Composition in Elderly
Brief Title: Motivational Resistance-training Program on Adherence and Body Composition in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Pablo Jorge Marcos Pardo, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PMAFI/03/12
Record Dates: First submitted 2017-06-19; First posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Motivation; Body Weight
Keywords: elderly; motivation; adherence; resistance-training; health
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Intervention Model Description: A quasi-experimental design (2x2) was developed, dividing the participants into two groups; one experimental and one control. In this design, an initial measurement prior to the intervention (pre-test) and a measurement after the intervention (post-test) were conducted. The sampling was natural and intentional.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- training group (Experimental): The training group, based on motivational strategies were performed and a moderate intensity training (8 to 12 repetitions). The load was increased: during the 12 weeks from 65% 1-RM to 80% 1-RM, performing individual more than the prescribed number of repetitions (12 repetitions). A 1-2 minutes resting period was allowed between sets. There was no attempt to control the velocity of the repetitions performed. Prior to each training session, the volunteers performed a specific warmup, consisting of 10 repetitions with approximately 50% of the load used in the first and second exercises of the training session. A total of 36 sessions were performed during the training period. This group was compared with no interventions subjects.
  Interventions: Other: Motivational resistance-training programme
- control group (No Intervention): The control group, did not participate in the motivational resistance-training program.

INTERVENTIONS:
Other: Motivational resistance-training programme — The experimental group exercised at a moderate intensity (8 to 12 repetitions). The load was increased during the 12 weeks from 65% 1-RM to 80% 1-RM. This training load was increased when the individual could perform more than the prescribed number of repetitions (12 repetitions), following the OMNI-RES scale and a hard effort perception level.74 A 1-2 minutes resting period was allowed between sets. During the sessions, the participants were verbally encouraged to perform the complete range of motion for each exercise and received motivational strategies.
  Arms: training group

SUMMARY:
Lack of physical activity is one of the major causes for obesity and functional disability in the elderly. Including regular exercise in elderly´s lifestyle is not an easy task. The main objective was to analyse the effect of a motivational resistance-training programme on satisfying the individual´s psychological needs, level of self-determination and body composition. A quasi-experimental study was performed with 47 volunteers (29 females, 18 males) of 67-75 years of age, divided into two groups: experimental (n = 27) and control (n = 20). A 12-week intervention programme was performed, with a total of 36 sessions.

DETAILED DESCRIPTION:
Material and Methods

Participants The study included a total of 47 subjects, (29 females, 18 males) ages 65 to 75 years, recruited from an elderly social club. The participants were divided into two groups: experimental group (n=27; 10 men and 17 female) and control group (n=20; 8 men and 12 female). The sampling was natural and intentional. All subjects originated from Murcia (Spain) and met the following inclusion criteria: had never previously attended classes in fitness academies or were not currently performing regular physical activity, and had no previous experience with resistance-training programmes. Exclusion criteria included any history of neuromuscular, metabolic, hormonal or cardiovascular diseases; not taking any medication that could influence hormonal and neuromuscular metabolism. In addition, the participants were advised to not alter their diet during the study. Participants were informed about the possible risks and discomforts that could arise and were asked to complete a health history questionnaire and sign a consent form. The current study was approved of the Ethics Committee of the Catholic University San Antonio of Murcia (Spain) following the guidelines of the Helsinki Declaration.

Design A quasi-experimental design (2x2) was developed, dividing the participants into two groups; one experimental and one control. In this design, an initial measurement prior to the intervention (pre-test) and a measurement after the intervention (post-test) were conducted. This same research design has been used in previous studies, which has sought to assess the effect of an intervention programme on body composition, motivational variables and resistance-training.

Data Collection and Procedure Motivational variables Behavioural regulation during exercise. The Spanish version of Behavioural Regulation during Exercise Questionnaire was used. This questionnaire allows to evaluate the type of motivational regulation related to physical exercise, and consists in 23 items distributed in three dimensions, based on the established distinction in the SDT between autonomous motivation, controlled motivation and demotivation. Autonomous motivation was calculated using the mean score of intrinsic regulation (e.g. "Because I think that exercise is fun"), integrated regulation (e.g. "Because I believe that physical exercise is consistent with my values") and identified regulation (e.g. "I value the benefits of exercise"). Each of these regulations was composed of 4 items, except for the identified regulations which was composed of 3 items. Controlled motivation was calculated using the mean score of introjected regulation (e.g. "I feel guilty when I don't exercise") and external regulation (e.g. "I feel under pressure from my friends/family to exercise") with 4 items each. Demotivation (e.g. "I don't see why I should have to exercise") was also calculated using 4 items. Previous research in the physical activity and health context demonstrated the internal reliability of the instrument.

Basic psychological needs during exercise. To assess the perceived need satisfaction of the participants, the Spanish adaptation of the Basic Psychological Needs in Exercise Scale was used (BPNES), which is specific for the context of physical activity and health.67 The questionnaire includes 12 items distributed in three dimensions. Four items measure autonomy (e.g. "I exercise according to what I intend to do"), four items measure competence (e.g. "I feel that physical exercise is an activity that I do very well") and the other four items measure relatedness (e.g. "I have a close relationship with the people with whom I exercise"). Previous research in the physical activity and health context demonstrated the internal reliability of the instrument.

The answers to the questionnaires were assessed on a Likert scale ranging from 1 to 7, where one corresponded with the anchor statement "strongly disagree" and seven with the anchor statement "strongly agree". Before carrying out the intervention, the main researcher contacted with the director of the social club to inform of the purpose of the study. Likewise, all the participants involved were informed about the process that they were going to follow, emphasizing that participation was voluntary. The researcher overviewed how to complete the questionnaire and answered any questions that arose during the process. The different questionnaires were completed in an adequate climate of concentration, with each participant taking approximately 15-20 minutes to complete the questionnaires.

Body composition variables Total body weight was measured, after removal of shoes and heavy outer clothing, using a Tanita BC-418 MA scale, (Tanita Corporation, Arlington Heights, IL) to the nearest 0.1 kg.69 Standing height without shoes was measured using a Seca 202 stadiometer (Seca, Hamburg, Germany) to the nearest 0.1 cm. To minimize the potential source of Bioimpedance systems (BIA) related to total body weight and height, body composition assessment was performed by a level two anthropometrist following International Society for the Advancement of Kinanthropometry recommendations.70 Body Mass Index (BMI) was calculated as the ratio of weight to squared height. BMI was categorized into underweight (<18.50 kg/m2), normal weight (18.50-24.99 kg/m2), overweight (25.00-29.99 kg/m2), and obese (30.00 kg/m2).

Bioelectrical impedance was measured using the Tanita BC-418 MA scale, with participants standing barefooted on the analyser's footpads, and holding its handles. Fat mass (FM) and muscle mass (MM) were then calculated, using the prediction equation described by Jebb et al. Bioelectrical impedance was chosen due to its ease of use and less invasive nature, making it suitable for assessment of body composition in vulnerable populations such as obese individuals and elderly.

Multi-dimensional intervention programme Prior to the commencement of the study, the subjects were submitted to two weeks of training, two sessions per week, in order to be familiarized with the resistance-training exercises performed in the current study. During this familiarization period, a higher emphasis was placed on learning the proper exercise techniques, and brief pauses between repetitions were allowed in order to reset their starting positions when necessary. During the second week of the familiarization period, a pre-test of the motivational variables was performed, as well as measuring weight, height, BMI, FM and MM. Both pre-test and post-test were carried out in one day between 8:00 and 9:00 a.m. After the pre-test, the experimental group underwent a resistance-training programme for 12 weeks, where different motivational strategies were used. The resistance-training programme incorporated resistance exercises of six major regions and consisted in 3 training sessions per week on non-consecutive days (Monday, Wednesday, and Friday). The six regions were chest, back, triceps, biceps, shoulders and legs. The different regions were grouped into a circuit. The control group, on the other hand, did not participate in the resistance-training programme.

The experimental group exercised at a moderate intensity (8 to 12 repetitions). The load was increased during the 12 weeks from 65% 1-RM to 80% 1-RM. This training load was increased when the individual could perform more than the prescribed number of repetitions (12 repetitions), following the OMNI-RES scale and a hard effort perception level. A 1-2 minutes resting period was allowed between sets.

All training sessions were monitored by an experienced physical education professional and the subjects were not allowed to perform any additional exercises during the training period. During the training weeks, participants were instructed not to change dietary habits or perform additional non-resistance-training related physical activity.

In addition, with the objective of increasing the adherence to the resistance-training programme, a series of motivational strategies were performed.

The strategies to motivation assessment used were based on the principles of the Self-Determination Theory (SDT). SDT includes a meta-theory for framing motivational studies, a formal theory that defines intrinsic and varied extrinsic sources of motivation, their role in cognitive and social development, as well as in individual differences. SDT is a theory of motivation and personality that addresses three universal, innate and basic psychological needs: autonomy, competence and relatedness. During the resistance-training programme, the subjects received verbal motivational strategies, based on previous studies which have proven the beneficial effect they exert on BPN satisfaction and autonomous motivation.

ELIGIBILITY:
Inclusion Criteria:

* Never previously attended classes in fitness academies or were not currently performing regular physical activity, and had no previous experience with resistance-training programmes

Exclusion Criteria:

* Any history of neuromuscular, metabolic, hormonal or cardiovascular diseases; not taking any medication that could influence hormonal and neuromuscular metabolism.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — older people
Enrollment: 47 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Change of behavioural regulation during exercise | Change from Baseline behavioural regulation during exercise at 12 weeks
  To evaluate the type of motivational regulation related to physical exercise. The Spanish version of Behavioural Regulation during Exercise Questionnaire was used. This questionnaire allows to 13 evaluate the type of motivational regulation related to physical exercise, and consists in 14 23 items distributed in three dimensions, based on the established distinction in the SDT 15 between autonomous motivation, controlled motivation and demotivation.
Change of basic psychological needs during exercise. | Change from Baseline Basic psychological needs during exercise at 12 weeks
  To assess the perceived need satisfaction of the participant. satisfaction of the participants, the Spanish adaptation of the Basic Psychological Needs 4 in Exercise Scale was used. The questionnaire includes 12 items distributed in three 6 dimensions.

SECONDARY OUTCOMES:
Change of body weight (kg) | Change from Baseline body weight (kg) at 12 weeks
  After removal of shoes and heavy outer clothing,using a Tanita BC-418 MA scale, (Tanita Corporation, Arlington Heights, IL) to the 24 nearest 0.1 kg
Change of standing height (cm) | Change from Baseline standing height (cm) at 12 weeks
  Assessed without shoes was measured using a Seca 202 stadiometer (Seca, Hamburg, Germany) to the nearest 0.1 cm.
Change of Body Mass Index (BMI): (kg/m^2) | Change from Baseline Body Mass Index (BMI): (kg/m^2) at 12 weeks
  was calculated as the ratio of weight to squared height
Change of bioelectrical impedance Muscle mass (kg) | Change from Baseline bioelectrical impedance Muscle mass (kg) at 12 weeks
  Was measured using the Tanita BC-418 MA scale, with participants standing barefooted on the analyser's footpads, and holding its handles.
Change of bioelectrical impedance Fat mass (%) | Change from Baseline bioelectrical impedance fat mass (kg) at 12 weeks
  Was measured using the Tanita BC-418 MA scale, with participants standing barefooted on the analyser's footpads, and holding its handles.

IPD SHARING:
Plan to Share IPD: No